CLINICAL TRIAL: NCT04425044
Title: Efficacy of AiM Covid Self Monitoring in Detecting Infection of COVID-19
Brief Title: AiM Covid Self Monitoring
Status: Completed | Type: Observational
Sponsor: Aarogyam UK (Other)
Collaborators: University of Warwick (Other); NMP Medical Research Institute (Other); Mothers Touch Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: Au015
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AiM Covid: Self Monitoring of symptoms in AiM Covid App
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — No Intervention

SUMMARY:
The objectives of this study are to test the level of accuracy of the prediction models that could be used as a 'digital test' to evaluate whether an individual is infected with COVID-19, based on their symptoms reported in the "AiM COVID-19" app

ELIGIBILITY:
Inclusion Criteria:

* Participants resident in India
* Voluntary completion of the self-test and evaluation.

Exclusion Criteria:

* People can not use mobile app
* Below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone worried about heath status relating with infection of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Fever | 1 day
  Self reported body temperature (Degrees Celsius)

SECONDARY OUTCOMES:
Shortness of Breath | 1 day
  Self reported shortness of breath symptom (tick box)
Cough | 1 day
  Self reported cough symptom (tick box)
Sore Throat | 1 day
  Self reported soar throat symptom (tick box)
Headache | 1 day
  Self reported headache symptom (tick box)
Muscle/ Joint Pain | 1 day
  Self reported muscle/ joint pain symptom (tick box)
Diarrhoea | 1 day
  Self reported diarrhoea symptom (tick box)
Vomiting/ Nausea | 1 day
  Self reported vomiting/ nausea symptom (tick box)
Runny Nose | 1 day
  Self reported runny nose symptom (tick box)
Loss of Smell/Taste | 1 day
  Self reported loss of smell/ taste symptom (tick box)
Other symptoms | 1 day
  Self reported other symptoms (tick box)

CONTACTS AND LOCATIONS:
Overall Officials: Vishwes Kulkarni, Principal Investigator — University of Warwick
Locations (2):
- India (2):
  - Mothers Touch Foundation, Mumbai, Maharashtra
  - NMP Medical Research Institite, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided